CLINICAL TRIAL: NCT06597916
Title: A Phase-2b Controlled Study to Evaluate the Humoral and Cellular Immune Response and Safety Following One and Two Doses of an Adjuvanted RSV Subunit Vaccine in Immunocompromised Patients Aged 18 Years and Older.
Brief Title: RSV Vaccination in Immunocompromised Patients.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Angelika Wagner, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ISPTM-RSV-001
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: RSV Infection
Keywords: RSV prophylaxis; RSV vaccine; RSV vaccination; RSV immunocompromised; RSV multiple myeloma; RSV lung cancer; RSV IBD
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Suspensions; Injections

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, parallel group, controlled, phase-2b
Who Masked: Participant
Masking Description: Controls will be randomized in a 1:1 ratio before study intervention at V1 to receive Arexvy / saline.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1-3 (2 times verum) (Experimental): Group 1-3 receive 2 doses of the RSV vaccine at visit 1 and visit 3, 1-2 months apart.
  Interventions: Biological: Arexvy powder and suspension for injection
- Group 4 (1 time verum, 1 time placebo, randomised) (Placebo Comparator): Group 4 receives 1 doses of the RSV vaccine or placebo at visit 1 and visit 3.
  Interventions: Biological: Arexvy powder and suspension for injection

INTERVENTIONS:
Biological: Arexvy powder and suspension for injection — Arexvy powder and suspension for injection (RSV vaccine)

SUMMARY:
Respiratory syncytial Virus (RSV) causes respiratory infections worldwide and typically presents with a seasonal pattern peaking in autumn/winter in temperate climate zones. Apart from infants and elderly individuals, patients with underlying substantial respiratory, cardiovascular, endocrinological diseases and immunocompromised patients are at increased risk to develop lower respiratory tract infection (LRTI) requiring intensive care associated with increased mortality. For certain risk groups such as patients after hematologic stem cell transplantation (HSCT) in-hospital mortality may be as high as 70 %. A causally related, RSV specific treatment does not exist and treatment is therefore usually supportive and non-specific.

The study is aiming to determine if immunocompromised patients benefit from two doses of a RSV subunit vaccine as opposed to one dose. The additional dose will be administered off label.

DETAILED DESCRIPTION:
The aim of this study is to assess immunogenicity and safety of the adjuvanted RSV vaccine Arexvy in different cohorts of immunocompromised patients. These data are needed as a basis for RSV vaccine recommendations.

Currently, one dose of the RSV vaccine is recommended for the elderly (≥ 60 years) according to the SmPC and national recommendations. However, it is not clear yet, whether in immunocompromised patients such as those with solid tumors, hemato-oncological malignancies with and without hematopoietic stem cell transplantation (HSCT) or those with biological treatments one dose of RSV vaccine would be sufficient to induce immune responses or if these patients would benefit from a second dose.

It is planned to evaluate immune responses after one and two doses with the adjuvanted RSV vaccine Arexvy in immunocompromised study groups compared to responses of healthy, elderly individuals receiving one vaccine dose only. Our analysis plan will include humoral and cellular immune responses after the first and second dose in immunocompromised patients belonging to different study groups compared to responses after one vaccine dose in controls.

ELIGIBILITY:
General inclusion criteria

1. Participants who, in the opinion of the investigator, can understand and will comply with the requirements of the protocol.
2. Participants living in the general community or in an assisted-living facility that provides minimal assistance can be enrolled, such that the participant is primarily responsible for self-care and activities of daily living.
3. Participants who can give written informed consent prior to study entry and performance of any study-specific procedure.
4. Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as hysterectomy, post-menopause, premenarche, bilateral oophorectomy, or bilateral salpingectomy
5. Female participants of childbearing potential may be enrolled in the study if the participant has practiced adequate contraception from 1 month prior to first Arexvy vaccination and agreed to continue adequate contraception for at least 1 month after completion of the last study intervention administration, and has a negative pregnancy test on the day of first vaccination prior to vaccine application.
6. Participants with chronic medical conditions with or without specific treatment are allowed to participate in this study if considered by the investigator as medically stable.
7. Additional inclusion criteria for "group 1":

   7.1. Age ≥18 years at the time of signing the Informed consent form (ICF). 7.2. Diagnosis of a hemato-oncological disease: multiple myeloma including early stage disease or lymphoma in participants medically stable in the opinion of the investigator at study inclusion.

   7.3. Participants without SCT or ≥3 months after autologous SCT until 24 months after SCT. SCT >24 months, if they have ongoing immunomodulatory/suppressive treatment.

   7.4. Immunosuppressive or modulating medication related to the hemato-oncological disease are allowed.
8. Additional inclusion criteria for "group 2":

   8.1. Age ≥18 years at the time of signing the Informed consent form (ICF). 8.2. Diagnosis of lung cancer ≥ stage 1. 8.3. Ongoing cancer treatment (including chemotherapy and immunotherapy) or initiation planned within 14 days and treatment initiation/vaccinations preferentially scheduled between treatment cycles.
9. Additional inclusion criteria for "group 3":

   9.1. Age ≥18 years at the time of signing the Informed consent form (ICF). 9.2. Diagnosis of an autoimmune/chronic inflammatory disease with chronic inflammatory bowel disease (IBD) or rheumatoid arthritis (RA).

   9.3. Treatment with biologicals such as TNF-alpha blocker, anti-CD20, JAK-inhibitors or other biological treatment (combinations with DMARDs, immunomodulators or steroidal or non-steroidal anti-inflammatory drugs are allowed).

   9.4. Stable disease at time of study entry.
10. Additional inclusion criteria for "group 4":

10.1. Age ≥60 years at the time of signing the Informed consent form (ICF). 10.2. Healthy, as established by medical history before entering the study with medically stable/controlled chronic conditions such as diabetes, hypertension or cardiac disease allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
To assess the mean geometric increase of RSV-A and RSV-B neutralizing antibodies after second vaccine dose over first vaccine dose with the adjuvanted RSV subunit vaccine Arexvy in immunocompromised patients ≥ 18 YoA. | up to 14 months per participant
  Fold increase of RSV-A and -B-specific neutralizing titers 30-60 days (V5) after the second dose relative to titers 30-60 days (V3) after the first dose in immunocompromised patients per group.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Specific Prophylaxis and Tropical Medicine, CePII, Medical university of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No